CLINICAL TRIAL: NCT01370746
Title: Perceived Barriers to Patient Adherence After Pediatric Solid Organ Transplantation (CTOTC-05)
Brief Title: Perceived Barriers to Patient Adherence After Pediatric Solid Organ Transplantation
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation in Children (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOTC-05
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Organ Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cross-Sectional Study Group: Cross-sectional comparison of perceived barriers to adherence to post-transplant immunosuppressant regimens in parents/legal guardians of children 0-11 years versus adolescents 12-21 years
- Longitudinal Study Group: Subset of Cross-Sectional Study Group to evaluate whether perceived barriers to adherence increase with time during the first year following transplantation

SUMMARY:
In this study, doctors will observe how and when pediatric patients who have received a solid organ transplant take their prescribed medication, and determining if there are reasons that keep these patients from taking all of their medicine.

DETAILED DESCRIPTION:
Adhering to treatment regimens after solid organ transplantation is critical for the prevention of complications, including acute and chronic organ rejection. It is important to recognize the perceived barriers to following treatment regimens and identify ways to address these barriers early in the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or guardian must be able to understand and provide informed consent/assent in English or Spanish
* Male or female primary solid organ transplant patients 0-21 years of age
* Recipients at least 1 month post-transplant hospital discharge

Exclusion Criteria:

* Inability or unwillingness of a participant or parent/guardian to give informed consent or comply with study protocol
* Condition or characteristic which in the opinion of the investigator makes the participant unlikely to complete the questionnaires
* Re-transplant recipient
* Multi-organ transplant recipient

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and pediatric patients after solid organ transplantation (heart, liver, or lung)
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Perceived barriers to adherence in adolescents and parent/legal guardian of pediatric patients | 1 month post transplant
  Barriers assessed using Brief Medication Questionnaire (BMQ); Adolescent Medication Barrier Scales questionnaire (AMBS); and Parent Medication Barriers Scale questionnaire (PMBS)
Change in perceived barriers to adherence from baseline to follow-up | 12 months post transplant
  Barriers assessed using Brief Medication Questionnaire (BMQ); Adolescent Medication Barrier Scales questionnaire (AMBS); and Parent Medication Barriers Scale questionnaire (PMBS)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Sweet, MD, PhD, Principal Investigator — Washington University School of Medicine; Lara Danziger-Isakov, MD, MPH, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - Ronald Reagan UCLA Medical Center (Mattel Childrens'), Los Angeles, California
  - University of California San Francisco Children's Hospital, San Francisco, California
  - Lucile Packard Children's Hospital at Stanford, Stanford, California
  - University of Florida Health Sciences Center, Gainesville, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Children's Hospital of Boston, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital of New York, New York, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - Children's Hospital and Regional Medical Center, Seattle, Washington

REFERENCES:
- [Background] Shemesh E. Barriers to adherence - To screen or not to screen, that is the question. Pediatr Transplant. 2016 Mar;20(2):188-90. doi: 10.1111/petr.12671. Epub 2016 Jan 22. No abstract available. PMID 26799519
- [Result] Danziger-Isakov L, Frazier TW, Worley S, Williams N, Shellmer D, Dharnidharka VR, Gupta NA, Ikle D, Sweet SC; CTOTC-05 Consortium. Perceived barriers to medication adherence in pediatric and adolescent solid organ transplantation. Pediatr Transplant. 2016 Mar;20(2):307-15. doi: 10.1111/petr.12648. Epub 2015 Dec 16. PMID 26670870
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Clinical Trials in Organ Transplantation in Children (CTOT-C) — https://www.ctotc.org/